CLINICAL TRIAL: NCT05541237
Title: Type 2 Diabetes Intervention by Gut Microbiota-directed Diet -a Open Labelled Randomized Controlled Trials
Brief Title: Type 2 Diabetes Intervention by Gut Microbiota-directed Diet -a Open Labelled RCT
Acronym: T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QiluH-T2D
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health (No Intervention)
- Disease (Experimental)
  Interventions: Dietary Supplement: Food

INTERVENTIONS:
Dietary Supplement: Food — Food
  Arms: Disease

SUMMARY:
This study is a randomized, open labelled, placebo-controlled clinical trial. The main purpose is to verify the superior effect of gut microbiota directed diet intervention over standard diet intervention by evaluating the changes of HbA1c relative to baseline at 16 weeks and 28 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes mellitus patients who have been diagnosed or screened for treatment without any hypoglycemic drugs;
* 6.5%≤HbA1c≤8.5%；
* FPG<10.0mmol/L;
* BMI≥24；

Exclusion Criteria:

* suspected other types of diabetes
* Moderate stroke occurred within one year;
* Frequent diarrhea or constipation in the past 3 months (more than 4 times / week);
* Acute complications occurred in the past 3 months, such as infection, ketosis and acidosis;
* Pregnant and lactating women (or women who are currently trying to conceive, or who are likely to have children and do not use contraceptives);
* Drinking (1 weeks of drinking more than 5 times, on average 2 two Baijiu or half Jin of yellow wine or 5 bottles of beer above);
* Those who have received drug treatment for the following diseases in the past three months: cholecystitis, peptic ulcer, urinary tract infection, acute pyelonephritis, cystitis, hyperthyroidism and other thyroid dysfunction;
* Gastrointestinal surgery (except appendicitis and hernia surgery);
* Antibiotics have been used in the past 3 months for 3 days or more;
* Physical methods, such as liposuction or gastrointestinal reconstruction, have been used to lose weight in the past 3 months;
* Physical disability, or inability to take care of themselves, recall and answer questions clearly due to other reasons;
* Anemia: hemoglobin < 10g / dl;
* Patients with severe liver diseases such as chronic hepatitis, persistent hepatitis and cirrhosis, and hepatitis B virus surface antigen (HBsAg) positive and abnormal liver function (serum alanine aminotransferase and aspartate aminotransferase are 2.5 times the normal value).
* Other serious diseases, such as malignant tumors, serious mental diseases, serious infectious diseases, etc;
* Patients who are participating in other intervention studies;
* In the judgment of the study physician, there are any conditions that affect the study compliance, such as:Alcohol or drug abuse in the past 12 months; Serious adverse drug treatment compliance in the past 12 months; The residence is far away from the research center, or it is planned to move far away or travel frequently in the next year; The clinical diagnosis of dementia or the judgment of cognitive function by the research physician will affect the research compliance; Other medical, psychological or behavioral factors that affect the study compliance are judged by the study physician.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-09-05 (Estimated); Study Completion 2024-09-08 (Estimated)

PRIMARY OUTCOMES:
changes of HbA1c compared with baseline | 28 weeks
  changes of HbA1c compared with baseline
remission rate | 28 weeks
  remission rate of T2D by ADA guideline；ratio of subjects whose blood glucose can reach completely normal without drug intervention

SECONDARY OUTCOMES:
control rate | at 16 weeks of treatment and 28 weeks of follow-up
  Proportion of subjects with HbA1c < 7.0%
blood lipid profile | at 16 weeks of treatment and 28 weeks of follow-up
  Changes of blood lipids (total cholesterol, triglyceride, high density lipoprotein cholesterol, low density lipoprotein cholesterol) relative to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China